CLINICAL TRIAL: NCT03023254
Title: An Exploratory Study to Assess the Efficacy of the Avène Hydrotherapy on Chronic Pruritus in Adults With Plaque Psoriasis
Brief Title: An Exploratory Study to Assess the Efficacy of the Avène Hydrotherapy
Acronym: PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PAP
Record Dates: First submitted 2016-10-25; First posted 2017-01-18 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pruritus Due to Plaque Psoriasis
MeSH Terms: interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrotherapy group (Other): Subjects included in the "hydrotherapy group" will undergo a 3-week Avène hydrotherapy in addition to their usual psoriasis and/or pruritus management (treatments and/or skin care products).
  Interventions: Other: Hydrotherapy
- Control group (No Intervention): Subjects included in the "control group" will not undergo the hydrotherapy and will keep following their usual psoriasis and/or pruritus management (treatments and/or skin care products).

INTERVENTIONS:
Other: Hydrotherapy — 3-week Avène hydrotherapy
  Arms: hydrotherapy group

SUMMARY:
To assess the benefit of the Avène hydrotherapy in subjects with pruritic plaque psoriasis

DETAILED DESCRIPTION:
* To assess the benefit of the Avène hydrotherapy in subjects with pruritic plaque psoriasis in the:

  * Improvement of pruritus
  * Improvement of psoriasis severity
  * Improvement of quality of life
  * Change of pruritus and psoriasis biological markers
  * Intake/application of treatments and skin care products for psoriasis and pruritus management, evaluated during a follow-up period
* To assess the time to pruritus relapse evaluated in subjects with pruritic plaque psoriasis, during the period following the Avène hydrotherapy (for the hydrotherapy group only)
* To assess the global efficacy of the Avène hydrotherapy in pruritic plaque psoriasis, according to subjects' and investigators' opinion (for the hydrotherapy group only)
* To assess the global cutaneous tolerance of the Avène hydrotherapy in subjects with pruritic plaque psoriasis (for the hydrotherapy group only)

ELIGIBILITY:
Inclusion Criteria:

* Subject with plaque psoriasis
* Subject with moderate to very severe chronic pruritus whose NRS score ≥ 4, (on a scale ranged from 0 to 10)
* Subject with chronic pruritus, i.e. for at least 6 weeks, due to plaque psoriasis

Exclusion Criteria:

* Subject with erythrodermic psoriasis, pustular psoriasis or palmoplantar keratoderma
* Subject with any other type of pruritus, not related to plaque psoriasis
* Subject with an acute, chronic or progressive disease other than plaque psoriasis which could be the origin of the pruritus
* Biotherapy, Phototherapy or PUVAtherapy treatment
* Psoriasis treatment by LASER
* Systemic or topical treatment taken/applied for psoriasis or pruritus management established or modified since the selection visit or planned to be established or modified between the inclusion visit and the end of the hydrotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Pruritus clinical criterion | Day18
  Pruritus intensity assessed by the subject on the NRS from 0 to 10

SECONDARY OUTCOMES:
Pruritus clinical criterion | Day1
  Pruritus intensity assessed by the subject on the NRS from 0 to 10
Pruritus clinical criterion | Day111
  Pruritus intensity assessed by the subject on the NRS from 0 to 10
Pruritus clinical criterion | Day202
  Pruritus intensity assessed by the subject on the NRS from 0 to 10
Psoriasis clinical criterion | Day1, Day18, Day111 and Day202
  Psoriasis Area Severity Index assessed by the investigator on a scale ranged from 0 to 72
Quality of life criterion | Day1, Day18, Day111 and Day202
  ItchyQoL questionnaire
Biological criterion (markers linked to neurogenic inflammation, epidermal differentiation, inflammation, antimicrobial peptides) | Day1, Day18, Day111 and Day202
  Psoriasis and pruritus biological markers
Hydrotherapy criterion | Day18
  Hydrotherapy global cutaneous tolerance on 4-point scale (0 = No effective ; 1=Little effective ; 2=Effective and 3=Very effective)

CONTACTS AND LOCATIONS:
Overall Officials: Diana PLACINTESCU, MD, Principal Investigator — Les Thermes d'Avène
Locations (29):
- France (27):
  - CHU Nord Service de Dermatologie, Amiens
  - CHU Angers Service de Dermatologie, Angers
  - Dr Martins-Hericher, Angers
  - CH de Boulogne sur Mer Hôpital DUCHENE - service de dermatologie, Boulogne-sur-Mer
  - CHU Morvan service de dermatologie, Brest
  - Dr Durbise, Cahors
  - Dr Parant, Clisson
  - Centre Hospitalier de Dunkerque - Service de Dermatologie, Dunkirk
  - Dr Abbadie, Langon
  - Dr Durieu, Lavaur
  - Dr Orsoni, Limoges
  - Dr Gutmann Heller, Lingolsheim
  - Dr Foucault, Lorient
  - Dr Nicol, Marseille
  - Dr Ruer-Mulard, Martigues
  - Hôpital St Eloi Service de Dermatologie, Montpellier
  - GHRMSA Hôpital Emile Muller Service de Dermatologie, Mulhouse
  - CHU Nantes - Unité Dermato-Cancérologie 7° nord Hotel Dieu, Nantes
  - Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD) - Hôpital l'Archet 2, Nice
  - CHU Nice - Hôpital l'Archet 1 - Centre de recherche clinique, Nice
  - Dr Fritsch, Obernai
  - Dr Pfister, Paris
  - CHU de Poitiers Pole régional de cancérologie Service de dermatologie, Poitiers
  - Centre hospitalier Poissy St germain, Saint-Germain-en-Laye
  - Dr Gadroy, Toulouse
  - CHRU Tours Service de Dermatologie, Tours
  - Dr Abdo-Morales, Tours
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau Dept. of Dermatology, Barcelona
  - Hospital Santa Caterina, Girona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thouvenin MD, Bacquey A, Babin M, Lestienne F, Lauze C, Gravier E, Placintescu D, Ortiz-Brugues A, Stander S. Efficacy of Avene Hydrotherapy on Chronic Pruritus in Patients with Plaque Psoriasis. Dermatol Ther (Heidelb). 2023 Dec;13(12):3137-3151. doi: 10.1007/s13555-023-01047-2. Epub 2023 Oct 14. PMID 37837493